CLINICAL TRIAL: NCT05296421
Title: Pilot Study to Investigate Targetable Metabolic Pathways Sustaining Pancreatic Cancer and Associated Genomic Alterations
Brief Title: Investigating Targetable Metabolic Pathways Sustaining Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Howard S. Hochster, MD, Associate Director for Clinical Research and Director, GI Oncology, Rutgers Cancer Institute, Director of Oncology Research, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 072107; NCI-2022-01787 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 072107; Pro2021001752 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Biopsy; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Basic science (uniformly-labeled [13C]glucose) (Experimental): Patients receive uniformly-labeled [13C]glucose IV over 10 minutes and then over up to 120 minutes until time of biopsy. Patients then undergo surgery and biopsy per standard of care.
  Interventions: Procedure: Biopsy; Procedure: Therapeutic Conventional Surgery; Other: Uniformly-labeled [13C]glucose

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Other: Uniformly-labeled [13C]glucose — Given IV
  Other Names: [U-13C] Glucose; U-13C-Glucose

SUMMARY:
This clinical trial investigates the nutrients pancreatic cancers depend on in which to survive and the processes these tumors use (metabolism) to obtain these nutrients. Giving U-13C-glucose during surgery may allow doctors to trace the metabolic activity of pancreatic cancer in research experiments done in the laboratory. These experiments may help researchers understand how cancer cells manage their nutrients when compared to normal pancreatic cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe and discover new insights into the glucose, tricarboxylic acid (TCA) cycle, amino acid, and lipid metabolic dependencies of pancreatic ductal adenocarcinoma (PDAC) via liquid chromatography-mass spectrometry (LC-MS) analysis of in vivo uniformly-labeled [13C]glucose (U-13C-glucose) labeled pancreatic cancer biopsies.

OUTLINE:

Patients receive uniformly-labeled [13C]glucose intravenously (IV) over 10 minutes and then over up to 120 minutes until time of biopsy. Patients then undergo surgery and biopsy per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >= 18 years of age
* Pancreatic adenocarcinoma patients, previously diagnosed by biopsy, who are candidates for intended curative resection either with or without neoadjuvant chemotherapy
* Willing to undergo mandatory intraoperative small excisional and core biopsies (4-6 passes) of tumor and normal tissue for research purposes at the time of proposed pancreatectomy
* 16 patients will be enrolled including 8 with no prior treatment and 8 treated with at least 3 months of neoadjuvant chemotherapy
* All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry

Exclusion Criteria:

* Patients receiving any anti-cancer therapy (chemotherapy, immunotherapy, and/or biologic therapy) for 8 patients; the other 8 patients will be treated with neoadjuvant chemotherapy but no radiation, biologic or immunotherapy prior to surgery
* Is currently enrolled, or will enroll in, a different clinical study in which investigational therapeutic procedures are performed or investigational therapies are administered while participating in this study
* Concomitant active malignancy
* Is of child-bearing potential who has not had a recent negative pregnancy test done outside of this clinical trial (i.e., as part of standard preparation for diagnosis and treatment for her cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
To measure glycolysis metabolism dependencies via liquid chromatography-mass spectrometry (LC-MS) | Up to 2 years
  To describe and discover new insights into the glucose metabolic dependencies of pancreatic ductal adenocarcinoma (PDAC) via liquid chromatography-mass spectrometry (LC-MS). The measure is to analyze in vivo U13C-glucose labeled pancreatic cancer biopsies. The blood collection will to allow for in depth evaluation of glycolysis metabolism

SECONDARY OUTCOMES:
To measure lipid metabolic dependencies via liquid chromatography-mass spectrometry (LC-MS) | Up to 2 years
  To describe and discover new insights into the lipid metabolic dependencies of pancreatic ductal adenocarcinoma (PDAC) via liquid chromatography-mass spectrometry (LC-MS) analysis of in vivo U13C-glucose labeled pancreatic cancer biopsies. The measure is to analyze in vivo U13C-glucose labeled pancreatic cancer biopsies. The blood collection will to allow for in depth evaluation of lipid metabolism

OTHER OUTCOMES:
To measure amino acid metabolism dependencies via liquid chromatography-mass spectrometry (LC-MS) | Up to 2 years
  To describe and discover new insights into the amino acid metabolic dependencies of Pancreatic ductal adenocarcinoma (PDAC) via liquid chromatography-mass spectrometry (LC-MS) analysis of in vivo U13C-glucose labeled pancreatic cancer biopsies. The measure is to analyze in vivo U13C-glucose labeled pancreatic cancer biopsies. The blood collection will to allow for in depth evaluation of amino acid metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Howard S Hochster, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Cooperman Barnabas Medical Center (Saint Barnabas Medical Center), Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No